CLINICAL TRIAL: NCT04865900
Title: Prevalence of Perimyocarditis After Covid-19 Vaccine
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: HYMC-0046-21
Record Dates: First submitted 2021-04-28; First posted 2021-04-29 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Perimyocarditis; Covid19
MeSH Terms: conditions — COVID-19 | interventions — Electrocardiography; Antibody Formation; Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Covid19 Vaccinated Patients: Patients who are planning to receive Pfizer-BioNTech BNT162b2 vaccines against Covid19
  Interventions: Diagnostic Test: Laboratory Blood Tests; Diagnostic Test: ECG; Diagnostic Test: PCR; Diagnostic Test: Antibody test; Diagnostic Test: Echocardiography; Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: Laboratory Blood Tests — Blood tests to determine liver and kidney functioning, total blood count, and troponin levels
Diagnostic Test: ECG — ECG to determine heart rate and functioning
Diagnostic Test: PCR — PCR test to determine whether patient has Covid19
Diagnostic Test: Antibody test — Antibody test to determine level of antibodies to Covid19
Diagnostic Test: Echocardiography — If Troponin level elevated echocardiography to determine heart function
Diagnostic Test: MRI — If Troponin level elevated MRI to determine heart function

SUMMARY:
The aim of this study is to determine whether there is a higher prevalence of perimyocarditis after undergoing vaccination for Covid-19.

ELIGIBILITY:
Inclusion Criteria:

* Patients planning Pfizer-BioNTech BNT162b2 vaccination against Covid19

Exclusion Criteria:

* Patients infected with Covid19

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patient Registries from local Health Maintenance Organizations
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-03-09 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Elevated Troponin | 4 weeks
  Laboratory blood tests will be taken before and after Covid19 vaccination and compared. Troponin levels above normal range of 0.4 ng/ml will indicate possibility of perimyocarditis and patient will referred for additional testing.

CONTACTS AND LOCATIONS:
Overall Officials: Saif Abu-Moch, MD, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel